CLINICAL TRIAL: NCT02302313
Title: Pilot Study of the ANI (Analgesia Nociception Index) Validity on the Nociception Assessment in Healthy Volunteers in State of Hypnosis, Compared to Painful Numerical Verbal Scale (EVN).
Brief Title: Study of the ANI Validity on Evaluation of Nociception in State of Hypnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: RB 13.186 ANI-HYPNOSE
Record Dates: First submitted 2014-09-10; First posted 2014-11-27 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: healthy volunteers; critical awareness; hypnosis; Analgesia Nociception Index; numerical verbal scale; Determine the validity of the index (ANI); nociception in critical awareness
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- painful stimuli (Other): No drug and no placebo will be used in this study. The study participants will only rate their pain on a numerical scale (EN) following cutaneous painful stimulation (6 for each phase) of variable intensity, delivered by a CO2 laser. ANI (Analgesia Nociception Index) will be raised simultaneously by the ANI monitor. This sequence will be performed on subjects at rest and in a state of hypnosis by the technique of "remembering a pleasant memory" and the ideo-sensory technique of "protective glove".
  Interventions: Device: CO2 laser and ANI monitor

INTERVENTIONS:
Device: CO2 laser and ANI monitor — Painful skin stimuli of variable intensity will be delivered by a CO2 laser used at the power of 0.3 W for each stimulation (6/phases) and this for each of the 3 phases (critical consciousness or hypnosis). During each stimulation, ANI values will be identified by the Physiodoloris ® monitor, through 3 standard ECG electrodes placed on the thorax of the subject.

SUMMARY:
Healthy subjects should assess pain on a numerical scale (EN), during painful skin stimuli of variable intensity delivered by a CO2 laser used at the power of 0.3 W, known for its safety. ANI (Analgesia Nociception Index) will be raised simultaneously. This sequence will be made on subjects at rest and in a state of hypnosis using the technique of "remembering a pleasant memory" and the ideo-sensory technique of "protective glove".

The average value of the ANI will be compared to the value of the EVN of pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* Knowledge of the state of hypnosis
* Healthy volunteers
* Capable adults
* Free and informed consent

Exclusion Criteria:

* Heart diseases
* Medication affecting the heart rate
* Medication affecting the skin sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
EVN value of pain intensity versus average value of the ANI | ANI average value : measured continuously for 60 seconds after the painful stimulation. EVN value : raised a few seconds after the painful stimulation
  ANI value (0 to 100, without unit of measure) recorded continuously for 60 seconds after the painful stimulation compared to the EVN value of the pain intensity, from zero to ten (numerical verval scale), and this for each of 6 painful stimuli intensities of each three consecutive phases of the study.

SECONDARY OUTCOMES:
EVN value of the arduousness of pain perception versus ANI value | ANI average value : measured continuously for 60 seconds after the painful stimulation. EVN value : raised a few seconds after the painful stimulation
  EVN value of the arduousness of pain perception, from zéro to ten, for a stimulation intensity, depending on the phase of the study, compared to the ANI.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé MUSELLEC, Principal Investigator — Saint-Gregoire Private Hospital Center
Locations (1):
- Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire, France